CLINICAL TRIAL: NCT07233239
Title: A Phase 1b, Multicenter, Open-Label, Single-arm Study to Evaluate the Efficacy and Safety of Cannabidiol Oral Solution (CBD-OS [GWP42003-P, JZP926]) in Participants Aged 12 to 75 Years for the Treatment of Focal-Onset Seizures
Brief Title: A Study to Evaluate the Efficacy and Safety of Cannabidiol Oral Solution (CBD-OS [GWP42003-P, JZP926]) for the Treatment of Focal-Onset Seizures
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Jazz Pharmaceuticals Research UK Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JZP926-105
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Focal Seizures
Keywords: Focal Seizures
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CBD-OS (Experimental): Participants who will receive open-label CBD-OS.
  Interventions: Drug: CBD-OS

INTERVENTIONS:
Drug: CBD-OS — Starting dose of CBD-OS will be administered as per the approved local product label
  Other Names: GWP42003-P; JZP926

SUMMARY:
Cannabidiol oral solution (CBD-OS) is approved in the US for the treatment of seizures associated with Lennox-Gastaut syndrome (LGS), Dravet syndrome (DS), or Tuberous sclerosis complex (TSC) in patients 1 year of age and older. This study will assess the efficacy and safety of CBD-OS in participants aged 12 to 75 years for the treatment of focal-onset seizures (FOS).

DETAILED DESCRIPTION:
This study will assess the efficacy of CBD-OS as an adjunctive treatment in reducing the frequency of focal seizures compared to baseline as well as the effect of CBD-OS on health outcome endpoints in early line and refractory participants with FOS. This study will also examine pharmacokinetics (PK), safety, and potential predictors or mediators of treatment response, including functional magnetic resonance imaging (fMRI) and neuropsychological testing in a substudy.

ELIGIBILITY:
Participants are eligible to be included in the main study only if all of the following criteria apply:

1. Participant has a documented diagnosis of focal epilepsy according to the ILAE Classification of Epilepsy, 2017, characterized by focal seizure types with typical interictal/ictal EEG findings (eg, focal sharp waves or slowing).
2. Participant is currently treated with at least 1, but no more than 4, antiseizure medications on a stable regimen.
3. Participant is aged 12 to 75 years old, inclusive, at Screening.

Participants are excluded from the study if any of the following criteria apply:

1. Has a concurrent, confirmed diagnosis of non-epileptic seizures or events that can confound the assessment of the efficacy measures, in the opinion of the investigator.
2. Has clinically significant unstable medical condition(s), other than epilepsy.
3. History of suicidal behavior, current suicidal risk as determined from history, or presence of active suicidal ideation as indicated by a positive response to Item 4 or Item 5 on the C-SSRS or is considered at risk of suicide or self-harm based on the clinical judgement of the investigator following interview with the participant and/or caregiver.
4. Has known or suspected hypersensitivity to cannabinoids or any of the excipients of the study intervention, such as sesame oil.
5. Is currently treated with Epidiolex or received treatment with Epidiolex within 28 days prior to Screening (Visit 1).
6. Is currently using or has used recreational or medicinal cannabis, cannabinoid/CBD based medications, products, or supplements (botanical or synthetic) within 28 days prior to Screening (Visit 1) and/or is unwilling to abstain for the duration of the study.
7. Presence of only nonmotor onset seizures or primary generalized epilepsies.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2027-11-29 (Estimated); Study Completion 2027-11-29 (Estimated)

PRIMARY OUTCOMES:
Percent change in countable focal seizure frequency compared to baseline | Baseline up to 16 weeks

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Banner University Medical Center-Phoenix, Phoenix, Arizona
  - UC San Diego, La Jolla, California
  - Yale University, New Haven, Connecticut
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Savannah Neurology Specialists, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Wayne State University, Detroit, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Hackensack Meridian Neuroscience Institute at JFK University Medical Center, Edison, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Boston Children's Health Physicians, Hawthorne, New York
  - Onsite Clinical Solutions, Charlotte, North Carolina
  - Velocity Clinical Research at Raleigh Neurology, Raleigh, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Cincinnati, Gardner Neuroscience Institute, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Child Neurology & Consultants of Austin, Austin, Texas
  - ANESC Research, El Paso, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - William S Middleton Memorial Veterans Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No